CLINICAL TRIAL: NCT07250763
Title: Optimization of Intravenous Unfractionated Heparin Starting Infusion Rate for Adult Patients With Deep Vein Thrombosis/Pulmonary Embolism or Cardiac Indications
Brief Title: Therapeutic Initial Heparin Dosing for Patients With Clots or Certain Heart Conditions Admitted to the Hospital
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U21-08-4517
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Atrial Fibrillation; Acute Cardiac Syndrome; Mechanical Heart Valve Recipients
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Retrospective chart review and data was used to develop a dosing equation that uses patient specific factors. Results of intervention group will be compared to the retrospective group.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- acute care patients prescribed heparin for treatment of DVT, PE or for conditions such as ACS, Afib (Experimental): This arm will be participants whose initial dose will be using the patient specific calculator
  Interventions: Drug: Initial Heparin Dose Modification

INTERVENTIONS:
Drug: Initial Heparin Dose Modification — A patient specific initial therapeutic dose calculator will be used to start the heparin drip. The aim is to start the patient on a dose that is or is close to the therapeutic dose - one that gets the patient to the goal outcome (lab value driven)
  Other Names: Use of a patient specific calculator to determine therapeutic dose at initiation of heparin

SUMMARY:
The goal of this clinical trial study is to test whether a mathematical calculation, using the patient's gender, weight and kidney function, can better predict a patient's heparin goal dose than a flat number of units per patient weight can. Participants will have the first dose of heparin infusion calculated, after which if adjustments are needed, the Hospital's prebuilt table for results driven dosing for this purpose is used. The researchers will compare the time it takes for the participants to get to the desired goal using the patient's information for calculation versus patients in the past who received the medication using the flat rate. The hypothesis is that the patients with enhanced personal data, gender, weight and kidney function, included for the initial dose, will get to their goal lab value sooner and with less chance of delay or overshooting the goal. A quicker time to goal lab value is beneficial to patients in many ways, including earlier treatment of the clot or coronary issue that the patient is experiencing.

DETAILED DESCRIPTION:
Heparin infusions are high-risk medications that must be titrated to effect within a narrow therapeutic anti-Xa range. Prolonging the time to reach the therapeutic range decreases the clinical effectiveness of the infusion and increases the potential for adverse drug events.

The intervention used in this study will be calculating the initial heparin infusion rates described below rather than dosing 18 units/kg/hr for the moderate-intensity protocol and 12 units/kg/hr with a dose cap of 1000 units/hr for the low-intensity protocol.

Moderate-Intensity Protocol (R2 = 0.48) Heparin infusion rate (unit/(kg*hr))=(1004.8-163.5*(1 if female)-4.8*(age in years)+14.6*(actual body weight in kg)-19.3*(BMI in kg/m^2))/(Actual body weight in kg)

Low-Intensity Protocol (R2 = 0.31) Heparin infusion rate (unit/(kg*hr))=(615.5-70.1*(1 if female)-1.7*(age in years)+10.1*(actual body weight in kg)-11.9*(BMI in kg/m^2))/(Actual body weight in kg)

All other components of heparin infusion management will be conducted per Inova Health System standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years-old
* Diagnosis by the attending physician with one of the following conditions for which anticoagulation with heparin in an Food & Drug Administration approved indication and considered the standard of care:
* Moderate-intensity anti-Xa protocol: new-onset deep vein thrombosis or pulmonary embolism, or mechanical heart valve
* Low-intensity anti-Xa protocol: atrial fibrillation, acute cardiac syndrome, embolic stroke
* Heparin infusion either has not started or has been initiated in the last 120 minutes

Exclusion Criteria:

* Use of extracorporeal membrane oxygenation or ventricular assist devices such as Impella pumps
* Diagnosis of thrombophilia/hypercoagulable state
* Concurrent use of direct-acting oral anticoagulants or low molecular weight heparins
* Baseline anti-Xa > 0.7
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with steady-state anti Xa level within goal range | up to 72 hours from infusion initiation
  The proportion of patients who have a heparin infusion charted as administered for at least 6 hours who achieve at least one steady state anti-Xa level in the goal range. A steady state anti-Xa level is defined as an anti-Xa level drawn a minimum of 6 hours since the last titration or bolus dose was charted as administered. The goal anti-Xa range is defined as 0.3 to 0.7 for the moderate-intensity protocol and 0.3 to 0.5 for the low-intensity protocol.

SECONDARY OUTCOMES:
Time to first anti-Xa level within goal therapeutic range | up to 72 hours from infusion initiation
  time from first heparin infusion administration to the first anti-Xa level within the therapeutic range. Therapeutic ranges are as defined to moderate and low intensity protocols. Variability across participants will be summarized using a standard deviation
Change in hemoglobin from baseline | baseline, through the study completion, an average of 5 days
  Absolute change in the measurement of the hemoglobin from start of the heparin infusion throughout the inpatient stay to see if the decrease is a delta of >2gm/dL. Events of >2g/dL will be summarized separately.
The Incidence of thrombosis during hospitalization | baseline, through the study completion, an average of 5 days
  Number of participants who experience thrombosis during hospitalization
Incidence of major bleeding events during hospitalization | baseline, through the study completion, an average of 5 days
  The number of participants who experience major bleeding events during hospitalization.
Length of stay in acute care setting | baseline, through the study completion, an average of 5 days
  Total duration of hospitalization in acute care setting in days
Mortality during hospitalization | baseline, through the study completion, an average of 5 days
  Proportion of participants who die from any cause during hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Alexandria Hospital, Alexandria, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in doing of Heparin Infusions. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The information will become available after publication acceptance has been received. This will be available from 6 months post publication and up to 24 months post publication date.
Access Criteria: Scientific researchers interested in the study information would need to contact the primary or sub investigator via email. The data requested will be reviewed by the internal research team, any necessary paperwork required at the time by the Inova research team will be shared with the requester. If appropriate paperwork is received by Inova, the data requested will be shared expeditiously

REFERENCES:
- [Background] Schurr JW, Muske AM, Stevens CA, Culbreth SE, Sylvester KW, Connors JM. Derivation and Validation of Age- and Body Mass Index-Adjusted Weight-Based Unfractionated Heparin Dosing. Clin Appl Thromb Hemost. 2019 Jan-Dec;25:1076029619833480. doi: 10.1177/1076029619833480. PMID 30841720
- [Background] Smythe MA, Priziola J, Dobesh PP, Wirth D, Cuker A, Wittkowsky AK. Guidance for the practical management of the heparin anticoagulants in the treatment of venous thromboembolism. J Thromb Thrombolysis. 2016 Jan;41(1):165-86. doi: 10.1007/s11239-015-1315-2. PMID 26780745
- [Background] Granger CB, Hirsch J, Califf RM, Col J, White HD, Betriu A, Woodlief LH, Lee KL, Bovill EG, Simes RJ, Topol EJ. Activated partial thromboplastin time and outcome after thrombolytic therapy for acute myocardial infarction: results from the GUSTO-I trial. Circulation. 1996 Mar 1;93(5):870-8. doi: 10.1161/01.cir.93.5.870. PMID 8598077
- [Background] Hirsh J, Raschke R, Warkentin TE, Dalen JE, Deykin D, Poller L. Heparin: mechanism of action, pharmacokinetics, dosing considerations, monitoring, efficacy, and safety. Chest. 1995 Oct;108(4 Suppl):258S-275S. doi: 10.1378/chest.108.4_supplement.258s. No abstract available. PMID 7555181
- [Background] Barletta JF, DeYoung JL, McAllen K, Baker R, Pendleton K. Limitations of a standardized weight-based nomogram for heparin dosing in patients with morbid obesity. Surg Obes Relat Dis. 2008 Nov-Dec;4(6):748-53. doi: 10.1016/j.soard.2008.03.005. Epub 2008 Jun 30. PMID 18586569
- [Background] Riney JN, Hollands JM, Smith JR, Deal EN. Identifying optimal initial infusion rates for unfractionated heparin in morbidly obese patients. Ann Pharmacother. 2010 Jul-Aug;44(7-8):1141-51. doi: 10.1345/aph.1P088. Epub 2010 Jun 29. PMID 20587743
- [Background] Fan J, John B, Tesdal E. Evaluation of heparin dosing based on adjusted body weight in obese patients. Am J Health Syst Pharm. 2016 Oct 1;73(19):1512-22. doi: 10.2146/ajhp150388. PMID 27646813
- [Background] Shlensky JA, Thurber KM, O'Meara JG, Ou NN, Osborn JL, Dierkhising RA, Mara KC, Bierle DM, Daniels PR. Unfractionated heparin infusion for treatment of venous thromboembolism based on actual body weight without dose capping. Vasc Med. 2020 Feb;25(1):47-54. doi: 10.1177/1358863X19875813. Epub 2019 Oct 18. PMID 31623539
- [Background] Zifko UA, Slomka PJ, Reid RH, Young GB, Remtulla H, Bolton CF. The cortical representation of somatosensory evoked potentials of the phrenic nerve. J Neurol Sci. 1996 Aug;139(2):197-202. PMID 8856653
- [Background] Raschke RA, Gollihare B, Peirce JC. The effectiveness of implementing the weight-based heparin nomogram as a practice guideline. Arch Intern Med. 1996 Aug 12-26;156(15):1645-9. PMID 8694662